CLINICAL TRIAL: NCT04768569
Title: Pharmaceutical Interventions for Noise-Induced Hearing Loss-Acute Exposure Treatment
Brief Title: Noise-Induced Hearing Loss-Acute Exposure Treatment
Acronym: PINIHL-AET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PINIHL Program terminated by DoD
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Texas (Other); Gateway Biotechnology, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PINIHL-AET
Record Dates: First submitted 2020-12-04; First posted 2021-02-24 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Hearing Loss, Noise-Induced
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — Zonisamide; Capsules; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blinded placebo-control trial with three parallel groups, to make use of a common control group.
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized in a balanced fashion into one of 3 arms: Zonisamide 100 mg pre-op, Placebo, or Zonisamide 100 mg post-op.
  To ensure double-blinding of the trial, each subject will be assigned a previously prepared envelope with one package labeled "1" and designated to be taken 4 hours prior to surgery and another package labeled "2" designated to be taken within 4-12 hours after surgery or when the patient is released clinically to oral medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Zonisamide Pre-op + Placebo Post-op (Active Comparator): For subjects randomized to zonisamide pre-op, the pre-op package will contain one zonisamide capsule (100 mg PO) and the post-op package will contain one placebo capsule that looks, smells, and tastes the same as zonisamide capsules.
  Interventions: Drug: Zonisamide 100Mg Cap; Drug: Placebo
- Placebo Pre-op + Placebo Post-op (Placebo Comparator): For the subjects randomized to placebo, both pre- and post-op packages will contain placebo capsules that looks, smells, and taste the same as zonisamide capsules.
  Interventions: Drug: Placebo
- Placebo Pre-op + Zonisamide Post-op (Active Comparator): For subjects randomized to zonisamide post-op, the pre-op package will contain one placebo capsule and the post-op package will contain one zonisamide capsule (100 mg PO).
  Interventions: Drug: Zonisamide 100Mg Cap; Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide 100Mg Cap — ZONEGRAN® is commercially available for oral administration as capsules containing 100 mg of Zonisamide.
  Other Names: Zonegran; ZNS
  Arms: Placebo Pre-op + Zonisamide Post-op; Zonisamide Pre-op + Placebo Post-op
Drug: Placebo — The placebo will contain microcrystalline cellulose which is the predominant filler in the generic capsule.
  Other Names: microcrystalline cellulose

SUMMARY:
The purpose of this study is to assess the safety and efficacy of zonisamide for the treatment of noise-induced hearing loss in adults.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded placebo-control trial with three parallel groups, to make use of a common control group. After being informed about the study expectations and potential risks, all individuals providing written informed consent will undergo screening to determine eligibility for study entry.

Participants who meet the eligibility requirements will be randomized in a balanced fashion into one of 3 arms:

Group 1) Zonisamide 100 milligrams (mg) pre-op + Placebo post-op; Group 2) Placebo pre- + placebo post-op; and Group 3) Zonisamide 100 mg post-op + placebo post-op

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo a skull-based surgery that requires at least 45 minutes of surgical-drilling
* At least 18 years of age
* Air conduction thresholds in the non-operated ears are to be no worse than 25 decibel (dB) hearing loss (HL) for pure tone average 0.5, 1, and 2 kilohertz (kHz) with no individual threshold greater than 30 dB HL, and no worse than 45dB HL at 4 kHz at screening.
* Observed air-bone gap < 10 dB HL at 0.5, 1, 2, and 4 kHz, with normal tympanometry.
* Ability to understand and willingness to sign an Institutional Review Board (IRB) approved written informed consent document.

Exclusion Criteria:

* History of known sulfa allergy or hypersensitivity to carbonic anhydrase inhibitors
* History of moderate-to-severe kidney or liver disease
* Acute viral, bacterial, fungal or parasitic infection
* History of seizures
* Currently pregnant or breast-feeding
* Any current or history of ear disorder and/or central auditory dysfunction in the non-operated ear
* History of ototoxic drug use
* Current use of strong/moderate 3A4 inhibitor/inducer and grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Buchman, MD, FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 participants were consented for the study and enrolled. However, after consent but before any study activities could occur (including randomization), one participant chose to no longer participate. This excluded participant did not complete any study activities after consent. Thus, only 23 participants were consented and completed study activities including randomization.
Period: Overall Study
Arm/Group | Zonisamide Pre-op + Placebo Post-op | Placebo Pre-op + Placebo Post-op | Placebo Pre-op + Zonisamide Post-op
Started | 8 | 7 | 8
Completed | 8 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide Pre-op + Placebo Post-op | Placebo Pre-op + Placebo Post-op | Placebo Pre-op + Zonisamide Post-op | Total
Number analyzed (Participants) | 8 | 7 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (15.2) | 49.7 (12.37) | 53.6 (9.75) | 51.0 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 6 | 17
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 7 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Ratio of PTS-positive Subjects
Description: The primary efficacy endpoint will be the proportion of PTS-positive subjects defined as the ratio of PTS-positive subjects to total number of subjects within each study arm/group. Subjects defined as PTS-positive will demonstrate an increase in threshold that is ≥10 dB HL at any frequency from 2-6 kHz post-surgery as compared to baseline audiogram.
Time Frame: 30 days
Population: ITT Sample Set
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide Pre-op + Placebo Post-op | Placebo Pre-op + Placebo Post-op | Placebo Pre-op + Zonisamide Post-op
Number analyzed (Participants) | 8 | 7 | 8
Participants
  PTS-positive Subjects at Post-op 30 Days Visit | 3 | 1 | 1
  PTS-negative Subjects at Post-op 30 Days Visit | 5 | 6 | 7

2. Secondary Outcome: The Rate of Distortion Product Otoacoustic Emissions (DPOAE) Shift
Description: The secondary efficacy outcome measures will be the rate of temporary cochlear change as measured by a DPOAE amplitude shift at any frequency that is significantly greater than the stability of each measurement (i.e., 95% confidence interval of each measurement do not overlap). The rate of DPOAE shift is the ratio of DPOAE shift-positive subjects to total subjects within each arm.
Time Frame: 30 days
Population: ITT Sample
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide Pre-op + Placebo Post-op | Placebo Pre-op + Placebo Post-op | Placebo Pre-op + Zonisamide Post-op
Number analyzed (Participants) | 8 | 7 | 8
Participants
  No shift | 2 | 2 | 1
  Shift | 4 | 4 | 1
  Excluded | 2 | 1 | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from time of oral dose at the surgery visit to the final visit (30 days post-op, +/- 3 days). Total period of time over which adverse event data were collected were 30 days +/- 3 days.
Arm/Group | Zonisamide Pre-op + Placebo Post-op | Placebo Pre-op + Placebo Post-op | Placebo Pre-op + Zonisamide Post-op
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/7 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide Pre-op + Placebo Post-op (N=8) | Placebo Pre-op + Placebo Post-op (N=7) | Placebo Pre-op + Zonisamide Post-op (N=8)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrial Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide Pre-op + Placebo Post-op (N=8) | Placebo Pre-op + Placebo Post-op (N=7) | Placebo Pre-op + Zonisamide Post-op (N=8)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Facial Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 7 (7)
Facial paresis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Long thoracic nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04768569/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT04768569/SAP_001.pdf